CLINICAL TRIAL: NCT02826239
Title: Evaluation of Postural Effects on Multiple-breath-washout Derived Lung Function Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-posture
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Healthy Controls; Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pulmonary healthy controls: patients without known pulmonary disease
  Interventions: Device: multiple breath washout test (MBW)
- pulmonary disease: patients with known or suspected pulmonary disease
  Interventions: Device: multiple breath washout test (MBW)

INTERVENTIONS:
Device: multiple breath washout test (MBW) — measured in upright and supine position

SUMMARY:
The investigators aim to evaluated the effect of postural changes on novel lung function parameters derived from multiple-breath-washout.

ELIGIBILITY:
Inclusion Criteria:

* patients with and without known pulmonary disease

Exclusion Criteria:

* pregnancy
* inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with and without known pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change of lung clearance index (LCI) as determined by multiple breath washout | 60 minutes

SECONDARY OUTCOMES:
repeatability of lung clearance index (LCI) | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No